CLINICAL TRIAL: NCT03631576
Title: CD123/CLL1 CAR-T Cell Therapy for Relapsed and Refractory Acute Myeloid Leukemia
Brief Title: CD123/CLL1 CAR-T Cells for R/R AML (STPHI_0001)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Jianda Hu, Director of the department of Hematology, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART-19-04
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Relapsed/Refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): CD123/CLL1 CAR-T Cells treat
  Interventions: Biological: CD123/CLL1 CAR-T Cells

INTERVENTIONS:
Biological: CD123/CLL1 CAR-T Cells — CD123/CLL1 CAR-T Cell Therapy

SUMMARY:
The treatment options for relapse/refractory B-cell acute myeloid leukemia(AML)are limited.CD123/CLL1 CAR-T Cells may have a permanent anti-tumor effect and became very attractive. This study aims to assess the safety and toxicity of CD123/CLL1 CAR-T Cells to patients with relapse/refractory AML.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Aged < 70 years
* Patients with relapsed/refractory AML
* Cardiac: Left ventricular ejection fraction ≥ 50%
* Adequate renal and hepatic function
* Performance status: Karnofsky ≥ 70%

Exclusion Criteria:

* Pregnant or lactating females.
* Any co-morbidity precluding the administration of CD123/CLL1 CAR-T Cells.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2021-08-10 (Estimated); Study Completion 2021-08-10 (Estimated)

PRIMARY OUTCOMES:
Leukemia free survival | 1 year

SECONDARY OUTCOMES:
Adverse events that are related to treatment | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China